CLINICAL TRIAL: NCT03297411
Title: Clinical Outcomes With Electroconvulsive Therapy: Insights From Computational Modelling
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Wesley Mission (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HC17286
Record Dates: First submitted 2017-09-14; First posted 2017-09-29 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: electroconvulsive therapy; computer modelling
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Each participant will be randomly allocated to a sequence of treatments using designs for crossover studies with fewer periods (3) than treatments (4) involving two sets of ECT electrode placements and two sets of pulse width.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and the outcome assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brief Temporoparietal ECT (Active Comparator): Brief Pulse Temporoparietal ECT
  Interventions: Procedure: Brief Temporoparietal ECT
- Ultrabrief Temporoparietal ECT (Active Comparator): Ultrabrief Pulse Temporoparietal ECT
  Interventions: Procedure: Ultrabrief Temporoparietal ECT
- Brief Frontoparietal ECT (Active Comparator): Brief Pulse Frontoparietal ECT
  Interventions: Procedure: Brief Frontoparietal ECT
- Ultrabrief Frontoparietal ECT (Active Comparator): Ultrabrief Pulse Frontoparietal ECT
  Interventions: Procedure: Ultrabrief Frontoparietal ECT

INTERVENTIONS:
Procedure: Brief Temporoparietal ECT — Electroconvulsive Therapy (Brief pulse width, Temporoparietal) The intervention in this study is different combinations of pulse width and ECT electrode placements.
  Arms: Brief Temporoparietal ECT
Procedure: Ultrabrief Temporoparietal ECT — Electroconvulsive Therapy (Ultrabrief pulse width, Temporoparietal) The intervention in this study is different combinations of pulse width and ECT electrode placements.
  Arms: Ultrabrief Temporoparietal ECT
Procedure: Brief Frontoparietal ECT — Electroconvulsive Therapy (Brief pulse width, Frontoparietal) The intervention in this study is different combinations of pulse width and ECT electrode placements.
  Arms: Brief Frontoparietal ECT
Procedure: Ultrabrief Frontoparietal ECT — Electroconvulsive Therapy (Ultrabrief pulse width, Frontoparietal) The intervention in this study is different combinations of pulse width and ECT electrode placements.
  Arms: Ultrabrief Frontoparietal ECT

SUMMARY:
This study will generate new information on how to optimise brain targets with ECT stimulation.

DETAILED DESCRIPTION:
This study will differentiate the brain regions which are related to the effectiveness of electroconvulsive therapy (ECT) as a treatment, from the brain regions associated with memory impairment, with ECT stimulation. This will be done by 1) testing effects on memory of 4 different forms of ECT, which stimulate the brain differently; 2) in a subset of participants, use computer modelling to assess the pattern of brain stimulation with the 4 forms of ECT, and match these results to memory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years; right-handed
* DSM-5 Major Depressive Episode
* Prescribed with a course of ECT

Exclusion Criteria:

* Diagnosis (as defined by DSM-V) of psychotic disorder (apart from Major Depressive Episode with Psychotic features), current drug or alcohol abuse or dependence;
* ECT treatments in last 3 months from a prior course of ECT;
* Score <23 on the Montreal Cognitive Assessment Battery (MoCA);
* Past or current neurological illness or injury, medical illness which may significantly affect neuropsychological function;
* Inability to give informed consent or comply with study procedures; or
* Not having worked or studied in an English speaking background (to ensure validity of neuropsychological testing).
* Not be claustrophobic (if having an MRI brain scan).
* Not have any metal in your head or body (if having an MRI brain scan).
* Likely non response to RUL forms of ECT, as indicated by past non response to RUL ECT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
HVLT-R | Approximately 30 min after ECT treatment
  Hopkins Verbal Learning Test-Revised
BVMT-R | Approximately 30 min after ECT treatment
  Brief Visual Memory Test-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, Principal Investigator — The University of New South Wales
Locations (1):
- Wesley Hospital Kogarah, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Martin DM, Alduraywish A, Bakir AA, Dokos PhD S, Bakouri M, Bai S, Sackeim HA, Loo CK. A Computational Modeling Study of Focal Electrically Administered Seizure Therapy and Frontoparietal Electroconvulsive Therapy. J ECT. 2025 Apr 3. doi: 10.1097/YCT.0000000000001135. Online ahead of print. PMID 40184538